CLINICAL TRIAL: NCT05686304
Title: Effectiveness of Internet-based Self-help Money Management Program in Increasing in Financial Self-efficacy Among the Adult Population With Severe Mental Illness: A Randomized Controlled Trial
Brief Title: Effectiveness of Internet-based Self-help Money Management Program Among Adult With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: Baptist Oi Kwan Social Service (Other)
Responsible Party: Principal Investigator, CHAN Ka Shing Kevin, Associate Professor, Head of Department of Psychology, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-2022-0425
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Severe Mental Illness
Keywords: Money Management Program
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Money management group (Experimental): Participants in the money management condition start the 4-week money management program immediately after randomization and complete the post-intervention assessment right after they finish the treatment. They will be invited to participate in an interview after completing the post-intervention assessment.
  Interventions: Behavioral: Internet-based self-help money management program
- Waitlist control group (No Intervention): Participants in the waitlist control group will wait for 4 weeks without the money management program and then complete the post-intervention assessment. The waitlist control participants will start a money management program (equivalent to that of the money management group) immediately after completing the post-intervention assessment.

INTERVENTIONS:
Behavioral: Internet-based self-help money management program — The online money management program course will consist of 4 weekly modules, incorporating the key components of money management and the Model of Human Occupation (MOHO), including the concept of money management, money management skill, and risk of financial exploitation.
  Arms: Money management group

SUMMARY:
This experimental study aims to develop an internet-based self-help money management program that improve financial self-efficacy and its associated adverse outcomes among adult population with severe mental illness. In particular, this study compares the efficacy of the internet-delivered self-help money management program with the wait-list control group.

The online money management program course will consist of 4 weekly modules, incorporating the key components of money management and the Model of Human Occupation (MOHO). The program include the concept of money management, money management skill, and risk of financial exploitation. The main component of each module will be presented in video format, quiz, and homework. Materials will be presented interactively to facilitate engagement.

DETAILED DESCRIPTION:
Money management is necessary for people with severe mental illness (SMI) to live safely in the community. Collective evidence has suggested that mental disorder leads to drift into poverty, is strong. Most of them struggle to meet basic needs with their existing income. Financial instability has been consistently linked to an increased risk of relapse. This experimental study aims to develop an internet-based self-help money management program that improve financial self-efficacy and its associated adverse outcomes among adult population with severe mental illness. Its efficacy will be compared with the wait-list control group. We hypothesized that (1) participants who received a money management program will improve financial self-efficacy after the intervention as compared with the wait-list controls; (2) participants from the money management program will have better financial well-being after the intervention as compared with the wait-list controls.

The online money management program course will consist of 4 weekly modules, incorporating the key components of money management and the Model of Human Occupation (MOHO), including the concept of money management, money management skill, and risk of financial exploitation. Each module will consist of the main component presented in video format, quiz, and homework. Materials will be presented interactively to facilitate engagement.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents
* Age ≥18 years
* Carrying a diagnosis of mental illness
* Being able to read Chinese
* Have a computer, tablet and/or smartphone device with Internet access
* Willing to give informed consent and comply with the trial protocol

Exclusion Criteria:

Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Assessment in Financial Self-Efficacy on the Financial Self-Efficacy Scale at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  The Financial Self-Efficacy Scale assess the change in a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Change from Baseline Assessment in Financial Behaviour at Post-Intervention Assessment and Follow-up Assessment | Before intervention, Immediately after intervention, and 4 weeks after intervention
  Change in financial behaviour is assessed by asking participants to indicate the extent to which they perform six positive financial behaviours in a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Change from Baseline Assessment in Financial Attitude at Post-Intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  Change in financial attitude is assessed by asking participants to indicate their views about performing six positive financial behaviours in a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Change from Baseline Assessment in Financial Well-Being on the CFPB Financial Well-Being Scale at Post-Intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The CFPB Financial Well-Being Scale assess the change in a 5-point Likert scale, ranging from 0 (not at all) to 4 (completely).

SECONDARY OUTCOMES:
Change from Baseline Assessment in Psychological Wellbeing on the World Health Organisation-Five Well-Being Index (WHO-5) at Post-Intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The WHO-5 assess the change in a 6-point Likert scale, ranging from 1 (at no time) to 6 (all of the time).
Change from Baseline Assessment in Anxiety Symptom on the General Anxiety Disorder-7 (GAD-7) at Post-Intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The GAD-7 assess the change in a 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day).
Change from Baseline Assessment in Depressive Symptom on the Patient Health Questionnaire-9 (PHQ-9) at Post-Intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The PHQ-9 assess the change in a 4-point Likert scale, ranging from 0 (not at all) to 3 (nearly every day).
Change from Baseline Assessment in Quality of Life on the Twelve-Item Short-Form (SF-12) Health Survey at Post-Intervention Assessment and Follow-up Assessment | Before intervention and Immediately after intervention, and 4 weeks after intervention
  The SF-12 assess the change in a combination of 5-point and 3-point Likert scale, ranging respectively from 1 (poor/ never) to 5 (excellent/ very much), and 1 (never) to 3 (very much).
Treatment adherence at the Interview after Post-Intervention Assessment | Immediately after Post-Intervention Assessment
  Treatment adherence is assessed by asking participants to report the number of sessions they had read, how long they had spent on the program, and how far they had followed the instructions.
Treatment satisfaction at the Interview after Post-Intervention Assessment | Immediately after Post-Intervention Assessment
  Treatment satisfaction is assessed by asking participants to report whether they like the treatment and whether they found it useful in a 10-point Likert scale, ranging from not at all suitable to very suitable.
Treatment satisfaction on the internet (Acceptability of the Internet for delivering online programs) at the Interview after Post-Intervention Assessment | Immediately after Post-Intervention Assessment
  Acceptability of the Internet for delivering online programs is assessed by asking participants to report how suitable, how convenient, how much they liked, and how worried they were about their privacy in a 10-point Likert scale, ranging from not at all suitable to very suitable.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin, Ka Shing CHAN, Principal Investigator — The Education University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Baptist Oi Kwan Social Service, Hong Kong
  - The Education University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No